CLINICAL TRIAL: NCT00133276
Title: Prophylactic Treatment of Peginterferon-associated Psychopathology. A Double-blind Placebo-controlled Trial on the Effects of Escitalopram (Lexapro®) in Patients Treated With Peginterferon and Ribavirin (POPS Study)
Brief Title: Prophylaxis of Psychiatric Symptoms During Anti-HCV Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Foundation for Liver Research (Other)
Responsible Party: Dr. R.J. de Knegt, Foundation for Liver Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HCV05-01
Record Dates: First submitted 2005-08-22; First posted 2005-08-23 (Estimated); Last update posted 2010-02-19 (Estimated); Status verified 2010-02

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Peg-interferon; Psychiatric side-effects
MeSH Terms: conditions — Hepatitis C | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Escitalopram
- 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Escitalopram — OD 5mg for 2 weeks; OD 10mg for 24 weeks; OD 5mg for 2 weeks
  Other Names: Lexapro
  Arms: 1
Other: Placebo
  Arms: 2

SUMMARY:
The treatment of chronic hepatitis C with peginterferon and ribavirin is highly effective but is hampered by peginterferon-induced psychopathology.

Prevention of peginterferon-induced psychopathology with selective serotonin reuptake inhibitors (SSRI's) (paroxetine) has been shown to be effective in patients treated with interferon for malignant disease. The aim is to study the effects of prophylactic treatment with escitalopram (another SSRI) on peginterferon-associated psychopathology in patients treated with peginterferon and ribavirin for chronic hepatitis C.

DETAILED DESCRIPTION:
The treatment of chronic hepatitis C with peginterferon and ribavirin is highly effective but is hampered by peginterferon-induced psychopathology.

Prevention of peginterferon-induced psychopathology with SSRI's (paroxetine) has been shown to be effective in patients treated with interferon for malignant disease. The aim is to study the effects of prophylactic treatment with escitalopram on peginterferon-associated psychopathology in patients treated with peginterferon and ribavirin for chronic hepatitis C.

Design: double blind, randomized controlled trial with two arms, maximum 40 patients per arm. Patients, starting with peginterferon and ribavirin, will be randomized to receive escitalopram therapy 10 mg per day (however, 5 mg in the first two weeks) or placebo.

Study population and selection: eighty patients receiving peginterferon alfa-2a (Pegasys 180 microgram) and ribavirin (Copegus 400 mg twice daily) will be included in the study.

Aims of the study:

1. to asses whether prophylactic treatment with escitalopram avoids significantly the occurrence of peginterferon-induced psychiatric disturbance; defined as an increase of two points on observer-based rating scales reflecting anxiety (BAS:BriefAnxietyScale), loss of concentration, depression and loss of impulse control (Montgomery and Asberg Depression Rating Scale: MADRS), and
2. to assess the frequency of major depression according to DSM IV criteria, in the escitalopram and placebo-treated patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 18-70 years of age
* Evidence of chronic hepatitis C by detectable serum HCV-DNA
* Hepatitis C genotype 1,2,3 or 4
* Indication for antiviral therapy of hepatitis C according to current clinical guidelines
* Written informed consent

Exclusion Criteria:

* History or other evidence of severe illness, malignancy or any other condition which would make the patient, in the opinion of the investigator, unsuitable for the study
* Abnormal thyroid stimulating hormone (TSH)
* Presence of contra-indications for antiviral therapy
* Concurrent psychiatric axis I diagnosis according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM IV) criteria, as the presence of a major depressive episode, bipolar disorder or psychotic disorder.
* Concurrent use of psychotropic drugs such as MAO-inhibitors, St John's wort, Lithium and 5 HT-agonists and antiepileptics.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-08; Primary Completion 2008-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of peginterferon-induced psychiatric disturbance

SECONDARY OUTCOMES:
Occurrence of major depression

CONTACTS AND LOCATIONS:
Overall Officials: Robert J De Knegt, MD, Principal Investigator — Erasmus MC University Hospital
Locations (3):
- Netherlands (3):
  - Erasmus MC University Hospital, Rotterdam, South Holland
  - AMC, Amsterdam
  - Radboud University Hospital, Nijmegen